CLINICAL TRIAL: NCT05053932
Title: Long-term Comparative Cerebrovascular Outcome After Transplantation vs Standard Care in Children With Sickle Cell Anemia ( DREPAGREFFE-2)
Brief Title: Long-term Comparative Cerebrovascular Outcome After Transplantation vs Standard Care in Sickle Cell Anemia
Acronym: DREPAGREFFE2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other); Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Other Study IDs: DREPAGREFFE2
Record Dates: First submitted 2021-05-12; First posted 2021-09-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Sickle Cell Disease; Cerebral Ischemia; Stenosis
Keywords: transplantation
MeSH Terms: conditions — Anemia, Sickle Cell; Brain Ischemia; Constriction, Pathologic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * One blood sample for the checking of anti-erythroid alloimmunisation and exposition of phosphatidyl-serine.
  * DNA and plasma will be frozen, stored for hypoxia-factors/angiogenesis and nitroso-redox stress analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients included in Drepagreffe 1 study (NCT01340404): biological collection
  Interventions: Other: blood collection

INTERVENTIONS:
Other: blood collection — blood collection

SUMMARY:
The purpose of the present observational study is to remotely reevaluate the cohort of 67 sickle cell patients with transcranial Doppler-detected cerebral vasculopathy included in the national "Sickle Cell Transplant" protocol and whose 1- and 3-year results were published in JAMA (Journal of the American Medical Association) in 2019 and in BHJ in 2020.

DETAILED DESCRIPTION:
The present observational study has the objective to reevaluate at distance the cohort of 67 children with sickle cell anemia enrolled in the "Drepagreffe"trial because of cerebral vasculopathy detected by transcranial Doppler. Results at 1 and 3 years were reported in JAMA in 2019 in BHJ in 2020. This trial was the first worldwide prospective study comparing transplantation to standard care in sickle cell disease. Velocities were highly significantly more reduced with a higher proportion of patients with normalized velocities and better quality of life after transplantation than on standard care. Despite a trend to a better ischemic lesions outcome at 3 years, the difference was not significant and cognitive performances were not different between both groups. The biologic study only assessed at enrollment and 1-year showed lower levels of Ang-2 and HGF (hepatocyte growth factor) after transplant and a significant and independent association between Doppler normalization probability with low Ang-2 and BDNF (brain-derived neurotrophic factor) levels.The aim of the present study is to reassess at 9-10 years this cohort with grants allowing to reevaluate cognitive functioning and hypoxia/angiogenic factors not realized in the systematic cohort follow-up

ELIGIBILITY:
Inclusion Criteria:

* Patient of legal age or minor who participated in the DREPAGREFFE research protocol [NCT 01340404] between December 2010 and June 2013,
* Having read and understood the information letter

Exclusion Criteria:

* Refusal to participate
* Patient deceased

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population concerned 67 patients included in 2011-2013 in the DREPAGREFFE protocol [NCT 01340404]
Sampling Method: Non-Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Long term evolution (at 9-10 years) of Ischemic lesion on brain magnetic resonance imaging 10-year measurement of ischemic lesion on magnetic resonance imaging | within 6 months of inclusion
  The MRI-scores, ranging from 0 (best outcome) to 10 (worst outcome), are obtained by adding up the ischemic lesion scores from the left and right sides, i.e., 3 for territorial or 2 for border zone (cortical and subcortical), 1 for white matter and 1 for basal ganglia infarcts and 0 if absent on each side.
Long term evolution (at 9-10 years) of arterial stenosis on cerebral and cervical magnetic resonance angiography | within 6 months of inclusion
  The MRA stenosis-scores, ranging from 0 (best outcome) to 32 (worst outcome) are defined as the weighted sums over the 8 assessed cerebral arteries, as 0 if no stenosis, 1 if mild stenosis (25-49%), 2 if moderate stenosis (50-74%), 3 if severe stenosis (75-99%), and 4 if occlusion.

SECONDARY OUTCOMES:
Long term evolution (at 9-10 years) of cognitive performance | within 6 months of inclusion
  Full Scale Intelligence Quotient (40= worst outcome, 160= best outcome) is measured by Wechsler Intelligence Scale for Children -Fourth Edition (WISC-4) for children 7-16 years of age and by WAIS-3 (Weschler Adult Intelligence Scale-3) for patients older than 16 years
Long term evolution (at 9-10 years) of quality of life | within 6 months of inclusion
  Quality of life assessment is collected using the French version of the Pediatric Quality of Life Inventory Generic Core Scale (PedsQLTM 4.0 generic core scales) (physical, emotional, social, school items) (0= worst outcome, 100= best outcome) via self-report and parent proxy-report
Evolution at 9-10 years of factors of hypoxia and oxidative stress | within 6 months of inclusion
  Assessment on plasma Phosphatidyl-serine expression VEGF, Angiopoietin-1 (Ang-1) and Angiopoietin-2 (Ang-2),EPO, HIF-1, BDNF, PDGF-AA

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - Hôpital Robert Debré AP-HP, Paris, IDF
  - Groupe hospitalier Pellegrin, Bordeaux
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Hôpital Henri Monr - APHP, Créteil
  - CHU de la Guadeloupe, La Guadeloupe
  - Hôpital Bicêtre AP-HP, Le Kremlin-Bicêtre
  - IHOPe, Lyon
  - CHU de Lyon, Lyon
  - Hôpital de la Timone, Marseille
  - CHU de Montpellier, Montpellier
  - Hôpital Necker - AP-HP, Paris
  - CH de Pau, Pau
  - CHU de Rennes, Rennes
  - Hôpital Hautepierre, Strasbourg

IPD SHARING:
Plan to Share IPD: No